CLINICAL TRIAL: NCT04314986
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study of AR882, a Potent Uricosuric Agent, in Healthy Adult Male Volunteers
Brief Title: Multiple Ascending Dose Study of AR882 in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arthrosi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: AR882-102
Record Dates: First submitted 2020-03-10; First posted 2020-03-19 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- AR882 (Dose A) (Experimental)
  Interventions: Drug: Cohort 1: AR882 or placebo
- AR882 (Dose B) (Experimental)
  Interventions: Drug: Cohort 2: AR882 or placebo
- AR882 (Dose C) (Experimental)
  Interventions: Drug: Cohort 3: AR882 or placebo
- AR882 (Dose D) (Experimental)
  Interventions: Drug: Cohort 4: AR882 or placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Cohort 1: AR882 or placebo; Drug: Cohort 2: AR882 or placebo; Drug: Cohort 3: AR882 or placebo; Drug: Cohort 4: AR882 or placebo

INTERVENTIONS:
Drug: Cohort 1: AR882 or placebo — AR882 or matching placebo administered once daily for 10 days
  Arms: AR882 (Dose A); Placebo
Drug: Cohort 2: AR882 or placebo — AR882 or matching placebo administered once daily for 10 days.
  Arms: AR882 (Dose B); Placebo
Drug: Cohort 3: AR882 or placebo — AR882 or matching placebo administered once daily for 10 days
  Arms: AR882 (Dose C); Placebo
Drug: Cohort 4: AR882 or placebo — AR882 or matching placebo administered once daily for 10 days
  Arms: AR882 (Dose D); Placebo

SUMMARY:
A study to assess multiple ascending doses of AR882 in healthy adult males.

ELIGIBILITY:
Inclusion Criteria:

* Screening serum uric acid level ≥ 4.5 mg/dL (268 µmol/L) and < 9 mg/dL (535 µmol/L)
* Body weight no less than 50 kg and body mass index (BMI) within the range of ≥18 and ≤33 kg/m2
* Must be free of any clinically significant disease that requires a physician's care and/or would interfere with study evaluations or procedures

Exclusion Criteria:

* Malignancy within 5 years, except for successfully treated basal or squamous cell carcinoma of the skin
* History of cardiac abnormalities
* History and/or presence of drug addiction or excessive use of alcohol

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety profile of AR882 based on incidence of adverse events | 22 Days
  Incidence of adverse events following multiple doses of AR882
To evaluate the safety profile of AR882 based on incidence of abnormal laboratory findings | 22 Days
  Incidence of abnormal laboratory findings following multiple doses of AR882
To evaluate the safety profile of AR882 based on incidence of abnormal electrocardiogram findings | 22 Days
  Incidence of abnormal electrocardiogram findings following multiple doses of AR882
To evaluate the safety profile of AR882 based on incidence of abnormal vital signs findings | 22 Days
  Incidence of abnormal vital signs findings following multiple doses of AR882
Area under the curve (AUC) for plasma AR882 | 15 Days
  Profile from plasma in terms of AUC following multiple doses of AR882
Time to maximum plasma concentration (Tmax) for AR882 | 15 Days
  Profile from plasma in terms of Tmax following multiple doses of AR882
Maximum plasma concentration (Cmax) for AR882 | 15 Days
  Profile from plasma in terms of Cmax following multiple doses of AR882
Apparent terminal half-life (t1/2) for AR882 | 15 Days
  Profile from plasma in terms of t1/2 following multiple doses of AR882
Amount excreted (Ae) into urine for AR882 | 15 Days
  Profile from urine in terms of Ae following multiple doses of AR882
Fractional Excretion (FEUA) for AR882 | 15 Days
  Profile from urine in terms of FEUA following multiple doses of AR882

SECONDARY OUTCOMES:
PD profile following multiple doses of AR882 | 15 Days
  Profile from serum uric acid concentrations over time

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty, Ltd., Melbourne, Victoria, Australia